CLINICAL TRIAL: NCT02030093
Title: Evaluation Study of the Effectiveness of a High- Versus Low-frequency Telephone-based and Sort Message-based (Sms) Continuing Care Provided to Patients Who Have Achieved a 12 Week In-patient Treatment for Alcohol Dependence
Brief Title: Telephone-Based Continuing Care for Alcohol Dependence
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 077/13
Record Dates: First submitted 2013-12-19; First posted 2014-01-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Telephone-based continuing care; Outcome monitoring
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- High-frequency telephone-based continuing care: High-frequency telephone-based continuing care
  Interventions: Behavioral: Telephone-based counseling
- Low-frequency telephone-based continuing care: Low-frequency telephone-based continuing care
  Interventions: Behavioral: Telephone-based counseling
- SMS group: SMS group
  Interventions: Behavioral: Telephone-based counseling
- Control group: Control group
  Interventions: Behavioral: Telephone-based counseling

INTERVENTIONS:
Behavioral: Telephone-based counseling — Telephone-based continuing care wil be provided to patients in different frequency

SUMMARY:
Alcohol dependency is the second most common psychiatric disorder and a major public health concern. As addictive disorders and now thought to be chronic disorders for many patients there is a need for the development of expanded treatment approaches. Because relapse is more often the rule than the exception the importance of continuing care after an initial phase of treatment is evident. Studies investigating telephone-based continuing care for patients with alcohol dependence have shown to be an effective form of step-down treatment after a previous stabilisation treatment program and provide extended recovery support. Therefore, the investigators hypothesize that alcohol abstinent patients who received high-frequency telephone-based or sms-based continuing care show significantly less relapses respectively more abstinent days six and twelve months after in-patient treatment compared to patients who receive low-frequency or no telephone-based continuing care.

DETAILED DESCRIPTION:
Background

Alcohol dependence is a major public health problem. Because of its relapsing nature of the disorder, alcohol and also drug dependence are now thought to be chronic disorders for many patients.Therefore, continuing care has become an important element in the treatment of alcohol dependence. Continuing care is referred to as ongoing care after an initial phase of intensive care and can be provided in different modalities and formats such as group counseling, telephone-based counseling, individual therapy and more. However, many substance-dependence patients do not attend any continuing care or abandon attending care to early. To approach this problem more flexible continuing care protocols that abstain from the traditional face-to-face counseling sessions have been developed to promote better adherence an improve disease management over time. Studies on continuing care revealed mixed results that depend on the duration of the intervention and the method of delivery services. Longer planned intervention and active approaches that bring the intervention to the patients seem to be more effective than traditional approaches in the management of addiction. For instance studies investigating telephone-based continuing care for patients with alcohol dependence have shown to be an effective form of step-dow treatment after a previous stabilisation treatment program and provide extended recovery support. Results revealed that telephone-based continuing care produced higher rates of abstinence than face-to-face standard continuing care, especially patient with low to moderate risk scores benefited therefrom. Furthermore, it is a feasible instrument to implement a low-budget follow-up system in routine outcome monitoring.

Objective

In this study, the investigators want to evaluate the effectiveness of a high- versus low-frequency telephone-based and a short message-based continuing care provided for patients who have achieved a 12 week in-patient treatment for alcohol dependence. The investigators hypothesize that telephone-based continuing care should help the patients to bridge the gap of an intensive in-patient treatment to out-patient environment and working life.

Methods

320 patients will be recruited through the Clinic Südhang (Bern) and the Forel Clinic (Zürich), both specialized clinics for treatment of alcohol dependency. Patients, age 18-65, will have attended a 12-week in-patient treatment program for alcohol dependency. Participants are divided in 4 groups (high-frequency-, low-frequency-, sms- and control- group) by randomization. Patients of the high-frequency and sms group will be contacted 9 times during the first 6 months while the low-frequency group will be called 2 times and the control group will not be contacted. All 4 groups are contacted after 6 months and 12 months. The telephone continuing care consists of several cognitive-behavioral therapy components and includes monitoring of substance use status and progress towards identified goals, identification of current and anticipated high risk situations as well as development and rehearsal of improved coping behaviors. Each call lasts approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependency
* 12-week in-patient treatment
* At least six month of abstinence after treatment
* Written informed consent

Exclusion Criteria

* Use of illegal drugs
* Continued in-patient treatment
* Cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the clinic Südhang (Bern) and the Forel clinic (Zürich), both specialized clinics for the treatment of alcohol dependency
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Number of days of alcohol abstinence | Six months

SECONDARY OUTCOMES:
Number of days of alcohol abstinence | One year

CONTACTS AND LOCATIONS:
Overall Officials: Leila Maria Soravia, Dr. phil., Study Chair — University of Bern
Locations (1):
- Dep. of Psychiatric Neurophysiology, Bern University Hospital, Bern, Switzerland